CLINICAL TRIAL: NCT05800327
Title: A Two-Stage Study of the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics and Immunogenicity of Various Doses of Levilimab When Administered Intravenously and Subcutaneously to Healthy Subjects and Subjects With Active Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-089-5/LUNAR
Record Dates: First submitted 2023-02-02; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Levilimab; Ilsira; anti-IL-6R; IL-6 receptor inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — levilimab

STUDY DESIGN:
Intervention Model Description: The study design assumes two sequential stages corresponding to Phase I and Phase III studies.
  Stage 1 This is an open-label, single-center, non-randomized cohort study of the safety and tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of single intravenous or subcutaneous levilimab injections administered to healthy subjects at ascending doses (modified 3+3 design).
  Stage 2 This is a randomized, comparative, double-blind, controlled clinical study to assess efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of levilimab when administered at repeated intravenous or subcutaneous doses in combination with methotrexate in subjects with active rheumatoid arthritis resistant to methotrexate monotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LVL162 group (Experimental): Levilimab 162 mg SC QW plus placebo starting from Week 0.
  Interventions: Drug: Levilimab
- LVL324 group (Experimental): Levilimab 324 mg SC Q2W plus placebo starting from Week 0.
  Interventions: Drug: Levilimab
- LVL648 group (Experimental): levilimab 648 mg IV Q4W plus placebo starting from Week 0.
  Interventions: Drug: Levilimab

INTERVENTIONS:
Drug: Levilimab — Subcutaneous or intravenous injection of levilimab with placebo.

SUMMARY:
This is a two-stage study of efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of various doses of levilimab when administered intravenously and subcutaneously to healthy subjects and subjects with active rheumatoid arthritis resistant to methotrexate monotherapy.

Aim of the Stage 1 is to study the tolerability, safety, immunogenicity, and main pharmacokinetic and pharmacodynamic parameters of levilimab after its single subcutaneous or intravenous administration at ascending doses to healthy subjects.

Aim of the Stage 2 is to confirm the efficacy and safety of levilimab 648 mg IV Q4W in combination with methotrexate and levilimab 324 mg SC Q2W in combination with methotrexate in subjects with active rheumatoid arthritis, resistant to methotrexate monotherapy.

DETAILED DESCRIPTION:
Stage 1: there are 3 dose levels and 5 cohorts. The subjects will be followed up for up to 71 days after the IP administration.

Stage 2: the main period of the study (Weeks 0-24) is blinded; study subjects will receive levilimab with placebo. At Week 24 the study will become open-label and all subjects will continue to receive levilimab. At week 28 patients who achieved the RA remission at week 24 will be switched to maintenance therapy of levilimab and will receive it through Week 52. Subjects who do not achieve remission at Week 24, will continue to receive levilimab from Week 28 to Week 52 inclusive corresponding to their treatment group.

ELIGIBILITY:
Inclusion Criteria (stage 1):

1. Signed Informed Consent Form for participation in the study.
2. Malegender.
3. Age 18-45 inclusive at the time of signing the ICF.
4. Healthy status confirmed by the history, physical examination, and laboratory parameters.
5. The absence of a history and signs of alcohol abuse or substance addiction at the time of signing the ICF, and a negative alcohol saliva screening test in combination with a negative urine drug test.
6. The ability of the subject to follow the Protocol procedures, according to the Investigator.
7. The readiness of the subject and their sexual partners with a childbearing potential to use reliable contraceptive measures from the date of signing the informed consent form throughout the study period and for 4 weeks after the administration of the investigational product. This requirement does not apply to the subjects and their partners who have undergone operative sterilization or the female partners of a subject who have been menopausal for more than 2 years.
8. Readiness not to drink alcohol within 24 hours prior to and 70 days after the administration of the investigational product.

Inclusion Criteria (stage 2):

1. Signed ICF for participation in the study.
2. Men and women aged ≥ 18 on the ICF signing day.
3. Rheumatoid arthritis that meets the ACR 2010 criteria, confirmed not less than 24 weeks before the ICF signing date. In the event that a subject has been diagnosed with rheumatoid arthritis in accordance with the ACR 1987 criteria, the physician-investigator must confirm the diagnosis in accordance with the ACR 2010 criteria during the screening period, with this information included in the primary documentation, if this has not been done previously and is not documented.
4. Methotrexate therapy during the 12 weeks prior to the ICF signing date.
5. Use of methotrexate at a stable dose during the 4 weeks prior to the ICF signing date (the methotrexate dose should be 15-25 mg per week, methotrexate dose of 10 mg may be used in case of intolerability/toxicity of a higher dose).
6. Failure of methotrexate when used over the 12 weeks before the ICF signing date (according to the Investigator).
7. Swollen joint count ≥ 6 (out of 66); tender joint count ≥ 6 (out of 68).
8. The presence of at least one of three criteria: 1) CRP ≥ 10 mg/L, 2) ESR ≥ 28 mm/h (Westergren method / capillary photometry), 3) morning stiffness that lasts longer than 45 minutes.
9. The ability of the subject to follow the Protocol procedures, according to the Investigator.
10. The readiness of the subject and their sexual partners with a childbearing potential to use reliable contraceptive measures from the date of signing the informed consent form throughout the study period and for 4 weeks after the administration of the last dose of the investigational product. This requirement does not apply to the subjects and their partners who have undergone operative sterilization or females who have been menopausal for more than 2 years.

Exclusion Criteria (Stage 1):

1. A history of treatment with the products containing monoclonal antibodies to interleukin 6 or its receptor.
2. A History of severe hypersensitivity reactions (angioneurotic edema, anaphylaxis, or multiple drug allergy).
3. Known allergy or intolerance to monoclonal antibody drugs (murine, chimeric, humanized, or fully human) or any other components of the investigational product.
4. Major surgery within 30 days before the signing of the ICF.
5. Severe infections (including those that required hospitalization or parenteral antibacterial, antiviral, antimycotic, or antiprotozoal agents) within 6 months before signing the ICF.
6. Use of systemic antibacterial, antiviral, antimycotic, or antiprotozoal agents within 2 months before signing the ICF.
7. More than 4 episodes of respiratory infections over the past 6 months before signing the ICF.
8. Impossibility to insert a venous catheter for blood sampling (for example, due to skin disease at venipuncture sites).
9. A history of fever over 40 °C.
10. A history of increased levels of hepatic transaminases above 2.5 x ULN.
11. Epileptic seizures, a history of seizures.
12. Depression, suicidal ideations/attempts at the screening or in the history.
13. Regular oral or parenteral administration of any medicinal products, including over-the-counter drugs, vitamins and dietary supplements, within less than 2 weeks before signing the ICF.
14. Use of medicinal products, including over-the-counter drugs, with a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) within 30 days before signing the ICF.
15. Use of medicinal products that affect the immune status (cytokines and their inducers, glucocorticoid hormones, etc.) within 2 months before signing the ICF.
16. BCG vaccination, vaccination with live attenuated vaccines and with any other vaccines within 12, 8 and 4 weeks before signing the ICF, respectively, as well as during screening.
17. Standard laboratory and investigation abnormalities.
18. Smoking over 10 cigarettes a day.
19. Consumption of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ L of beer, 200 mL of wine or 50 mL of spirits) or a history of alcoholism, drug addiction, or drug abuse.
20. Donation of 450 mL or more of blood or plasma within 2 months prior to signing the ICF.
21. Participation in clinical trials of medicinal products within 2 months before signing the ICF or concurrent participation in other clinical trials.
22. Previous participation in the same clinical trial (excluding subjects who dropped out at screening and did not receive the IP).

Exclusion Criteria (Stage 2):

1. Previous exposure to tocilizumab or other monoclonal antibodies to the interleukin 6 / interleukin 6 receptor.
2. Previous therapy with Janus kinase inhibitors.
3. Previous exposure to rituximab or other products that cause depletion or suppression of B cell activity.
4. Felty's syndrome (regardless of form).
5. The functional status of the subject is class IV according to the ACR 1991 classification.
6. Known allergy or intolerance to any component of the study drug.
7. Concomitant treatment with the following products:

   * the need for prednisolone or its equivalent at an oral dose of more than 10 mg/day;
   * the need for oral prednisolone or its equivalent at a dose of ≤10 mg/day if this dose was not stable during the last 4 weeks before signing the ICF (patients who received topical glucocorticoids can be included in the study);
   * the need for NSAID use if the NSAID dose was not stable during the last 4 weeks before signing the ICF (the patients who occasionally received NSAIDs for fever or allergic syndrome in case of intercurrent diseases can be included);
   * the use of alkylating agents at any time within 12 months before signing the ICF;
   * intra-articular administration of glucocorticoids within 4 weeks before signing the ICF;
   * vaccination with live or attenuated vaccines at any time within 8 weeks before signing the ICF;
   * the use of leflunomide within 8 weeks before signing the ICF;
   * therapy with TNF-α inhibitors or T cell co-stimulation blockers within 8 weeks before signing the ICF.
8. Patients with any of the following laboratory findings at screening:

   * the content of hemoglobin in the blood < 80 g/L;
   * the number of leukocytes in the blood < 3.0 × 109/L;
   * the number of platelets in the blood < 100 × 109/L;
   * the number of neutrophils in the blood < 2 × 109/L;
   * AST and ALT levels ≥ 1.5 × ULN approved in the laboratory;
   * serum creatinine ≥ 1.7 × ULN approved in the laboratory.
9. Positive pregnancy urine test in women at screening (the test is not performed in women who have been menopausal for at least 2 years or who have undergone operative sterilization; any of these conditions must be documented).
10. A confirmed diagnosis or a history of the severe immunodeficiency of any other nature.
11. Diagnosis of HIV infection, hepatitis B, C.
12. Diagnosis of tuberculosis, including a history of tuberculosis.
13. Latent forms of tuberculosis (positive Diaskintest® or positive result of the QuantiFERON®-TB Gold test or T-SPOT.TB test, in the absence of radiographic signs of pulmonary tuberculosis).
14. A history of or current herpes zoster.
15. Documented chickenpox within less than 30 days before signing the ICF.
16. The confirmed diagnosis of another chronic infection (for example, invasive mycoses, histoplasmosis, etc.), which can increase the risk of infectious complications in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety primary endpoint (Stage 1) | Up to day 71
  To determine the safety profile of levilimab following its single subcutaneous or intravenous administration at ascending doses in healthy subjects.
Low disease activity (Stage 2) | Up to Week 24
  Proportion of subjects with low activity of rheumatoid arthritis (DAS28-ESR <3.2) at Week 24 of the study in each treatment group.

SECONDARY OUTCOMES:
RA remission (Stage 2, main period) | Up to Week 24
  Proportion of subjects who achieved RA remission according to DAS28-CRP (<2.6), DAS28-ESR (<2.6), CDAI (≤2.8), SDAI (≤3.3), and ACR/EULAR 2011
RA remission (Stage 2, main period) | Up to Week 52
  Proportion of subjects who achieved RA remission according to DAS28-CRP (<2.6), DAS28-ESR (<2.6), CDAI (≤2.8), SDAI (≤3.3), and ACR/EULAR 2011
PK endpoints (Stage 1) | Up to Week 52
  AUC0-1680
PK endpoints (Stage 1) | Up to Week 24
  AUC0-1680
PK endpoints (Stage 1) | Up to Week 24
  AUC0-∞
PK endpoints (Stage 1) | Up to Week 52
  AUC0-∞
PK endpoints (Stage 1) | Up to Week 24
  Cmax
PK endpoints (Stage 1) | Up to Week 52
  Cmax
PK endpoints (Stage 1) | Up to Week 24
  Cmin
PK endpoints (Stage 1) | Up to Week 52
  Cmin
PK endpoints (Stage 1) | Up to Week 24
  Tmax
PK endpoints (Stage 1) | Up to Week 52
  Tmax
PK endpoints (Stage 1) | Up to Week 24
  Tmin
PK endpoints (Stage 1) | Up to Week 52
  Tmin
PK endpoints (Stage 1) | Up to Week 24
  Vd
PK endpoints (Stage 1) | Up to Week 52
  Vd
PK endpoints (Stage 1) | Up to Week 24
  T½
PK endpoints (Stage 1) | Up to Week 52
  T½
PK endpoints (Stage 1) | Up to Week 24
  Kel
PK endpoints (Stage 1) | Up to Week 52
  Kel
PK endpoints (Stage 1) | Up to Week 24
  CL
PK endpoints (Stage 1) | Up to Week 52
  CL
ACR response (Stage 2, main period) | Week 24, 52
  Proportion of subjects who achieved ACR20, ACR50 and ACR70
Low disease activity (Stage 2, main period) | Week 24, 52
  Proportion of subjects with low rheumatoid arthritis activity according to DAS28-CRP (<3.2), DAS28-ESR (<3.2), CDAI (≤10), SDAI (≤11)
Changes in RA indexes (Stage 2, main period) | Week 24, 52
  Change in DAS28-CRP, DAS28-ESR, CDAI and SDAI from baseline
Moderate/good response according to the EULAR criteria (Stage 2) | Week 24, 52
  Proportion of subjects with moderate and good response according to the EULAR criteria at Week 24 and 52 compared with baseline values.
Change in the serum C-reactive protein concentration (Stage 2) | Week 24, 52
  Change in the serum C-reactive protein concentration from baseline
Change in ESR (Stage 2) | Week 24, 52
  Change in ESR from baseline
Change in the quality of life measured with SF-36 (Stage 2) | Week 24, 52
  Change in the quality of life according to the SF-36 questionnaire from baseline
Change in the quality of life measured with the EQ-5D-3L (Stage 2) | Week 24, 52
  Change in the quality of life according to the EQ-5D-3L questionnaire from baseline
Change in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score (Stage 2) | Week 24, 52
  Change in the fatigue assessments according to the FACIT-F questionnaire from baseline
Change in functional activity (Stage 2) | Week 24, 52
  Change in the functional activity according to the HAQ-DI questionnaire from baseline
X-Ray assessment (Stage 2) | Week 24, 52
  Radiographic characterization of the affected joints at Week 24: change in mean modified total Sharp/van der Heijde score (mTSS).
Key Secondary PK endpoint (Stage 2) | Week 24
  Ctrough geometric mean in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- X7 Clinical Research, Saint Petersburg, Russia

REFERENCES:
- [Result] Lomakin NV, Bakirov BA, Protsenko DN, Mazurov VI, Musaev GH, Moiseeva OM, Pasechnik ES, Popov VV, Smolyarchuk EA, Gordeev IG, Gilyarov MY, Fomina DS, Seleznev AI, Linkova YN, Dokukina EA, Eremeeva AV, Pukhtinskaia PS, Morozova MA, Zinkina-Orikhan AV, Lutckii AA. The efficacy and safety of levilimab in severely ill COVID-19 patients not requiring mechanical ventilation: results of a multicenter randomized double-blind placebo-controlled phase III CORONA clinical study. Inflamm Res. 2021 Dec;70(10-12):1233-1246. doi: 10.1007/s00011-021-01507-5. Epub 2021 Sep 29. PMID 34586459